CLINICAL TRIAL: NCT03751072
Title: Efficacy and Toxicity of Blinatumomab in the French Compassionate Use Program (ATU) for Adult Patients With B-cell Precursor Acute Lymphoblastic Leukemia (BCP-ALL) Refractory, in Relapse, or With Positive Minimal Residual Disease.
Brief Title: Efficacy and Toxicity of Blinatumomab in the French ATU for Adult BCP-ALL R/R, or With MRD+ (FRENCH-CYTO)
Acronym: FRENCH-CYTO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Group for Research in Adult Acute Lymphoblastic Leukemia (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: FRENCH-CYTO
Record Dates: First submitted 2018-10-11; First posted 2018-11-23 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Acute Lymphoblastic Leukemia, in Relapse; Acute Lymphoblastic Leukemia With Failed Remission
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Relapse/Refractory
- MRD positive

SUMMARY:
The outcome of young adults (18-60 years) with ALL has been dramatically improved by the use of pediatric-inspired trials. About 60% of these young adult patients will be cured at 5 years. In this context, early evaluation of minimal residual disease (MRD) at complete remission has been shown to be one of the most powerful prognostic factor, but also predictive of the benefit of allogeneic stem cell transplantation (ASCT). Despite this global improvement, about 30% of patients experience a relapse and will be exposed to be refractory to salvage therapy or to early disease escape. In adult ALL, the most important prognostic factors at relapse are : the time from first CR to relapse, the achievement of a second complete remission (CR), and the feasibility of ASCT.

Blinatumomab is a bispecific T-cell engager that recruits T-cell on CD19 positive blast cells and induces anti-leukemic cytotoxicity. In a phase 3 trial in relapse/refractory Philadelphia-negative (Ph-) ALL, 43% of patients achieved a CR or CR with partial hematological recovery (CRh), with the majority of responses occurring within the first cycle. In patients with positive MRD (MRD+) BCP-ALL, blinatumomab resulted in complete MRD response in 78% of patients after one cycle.

Between 2012 and 2016, blinatumomab was available in France for R/R and MRD+ ALL adult patients through the French Compassionate Use Program. About 92 adult ALL were treated at different stages of the disease in 27 centers.

DETAILED DESCRIPTION:
To evaluate the efficacy of blinatumomab given in the French Compassionate Use Program, in term of overall survival in both R/R (first cohort) and MRD positive (second cohort) patients.

To evaluate the efficacy of blinatumomab given in the French Compassionate Use Program, in term of CR/CRH in R/R patients, To evaluate the efficacy in term of molecular response in both R/R and MRD+ cohorts, To evaluate the efficacy of blinatumomab given in the French Compassionate Use Program, in both Ph+/Ph- ALL patients To evaluate the feasibility and the safety of blinatumomab administration in a multi-center setting.To evaluate the feasibility of allogeneic stem cell transplant after blinatumomab administration in both populations.

ELIGIBILITY:
Inclusion Criteria:

Patient with Philadelphia-negative or positive (Ph+) ALL in relapse, refractory to salvage therapy, or with MRD positive ALL that received blinatumomab in the French ATU program.,

* Patient treated in the GRAALL network,
* Patient who does'nt object to participate in the study

Exclusion Criteria :

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients aged 18y+ with R/R or MRD+ BCP-ALL treated in the French GRAALL Network
Sampling Method: Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2018-07-16 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2019-01-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival in R/R and MRD+ cohorts | 6 months
  Months

SECONDARY OUTCOMES:
Response rates | 6 months
  Percent
Adverse events | 6 months
  Percent
Disease free survival | 6 months
  Months

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas BOISSEL, MD, Principal Investigator — 142499643
Locations (1):
- CABANNES-HAMY Aurélie, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dombret H, Cluzeau T, Huguet F, Boissel N. Pediatric-like therapy for adults with ALL. Curr Hematol Malig Rep. 2014 Jun;9(2):158-64. doi: 10.1007/s11899-014-0210-9. PMID 24682859
- [Background] Dhedin N, Huynh A, Maury S, Tabrizi R, Beldjord K, Asnafi V, Thomas X, Chevallier P, Nguyen S, Coiteux V, Bourhis JH, Hichri Y, Escoffre-Barbe M, Reman O, Graux C, Chalandon Y, Blaise D, Schanz U, Lheritier V, Cahn JY, Dombret H, Ifrah N; GRAALL group. Role of allogeneic stem cell transplantation in adult patients with Ph-negative acute lymphoblastic leukemia. Blood. 2015 Apr 16;125(16):2486-96; quiz 2586. doi: 10.1182/blood-2014-09-599894. Epub 2015 Jan 13. PMID 25587040
- [Background] Gokbuget N, Stanze D, Beck J, Diedrich H, Horst HA, Huttmann A, Kobbe G, Kreuzer KA, Leimer L, Reichle A, Schaich M, Schwartz S, Serve H, Starck M, Stelljes M, Stuhlmann R, Viardot A, Wendelin K, Freund M, Hoelzer D; German Multicenter Study Group for Adult Acute Lymphoblastic Leukemia. Outcome of relapsed adult lymphoblastic leukemia depends on response to salvage chemotherapy, prognostic factors, and performance of stem cell transplantation. Blood. 2012 Sep 6;120(10):2032-41. doi: 10.1182/blood-2011-12-399287. Epub 2012 Apr 4. PMID 22493293
- [Background] Topp MS, Gokbuget N, Stein AS, Zugmaier G, O'Brien S, Bargou RC, Dombret H, Fielding AK, Heffner L, Larson RA, Neumann S, Foa R, Litzow M, Ribera JM, Rambaldi A, Schiller G, Bruggemann M, Horst HA, Holland C, Jia C, Maniar T, Huber B, Nagorsen D, Forman SJ, Kantarjian HM. Safety and activity of blinatumomab for adult patients with relapsed or refractory B-precursor acute lymphoblastic leukaemia: a multicentre, single-arm, phase 2 study. Lancet Oncol. 2015 Jan;16(1):57-66. doi: 10.1016/S1470-2045(14)71170-2. Epub 2014 Dec 16. PMID 25524800
- [Background] Gokbuget N, Dombret H, Bonifacio M, Reichle A, Graux C, Faul C, Diedrich H, Topp MS, Bruggemann M, Horst HA, Havelange V, Stieglmaier J, Wessels H, Haddad V, Benjamin JE, Zugmaier G, Nagorsen D, Bargou RC. Blinatumomab for minimal residual disease in adults with B-cell precursor acute lymphoblastic leukemia. Blood. 2018 Apr 5;131(14):1522-1531. doi: 10.1182/blood-2017-08-798322. Epub 2018 Jan 22. PMID 29358182
- [Background] Lee DW, Gardner R, Porter DL, Louis CU, Ahmed N, Jensen M, Grupp SA, Mackall CL. Current concepts in the diagnosis and management of cytokine release syndrome. Blood. 2014 Jul 10;124(2):188-95. doi: 10.1182/blood-2014-05-552729. Epub 2014 May 29. PMID 24876563